CLINICAL TRIAL: NCT05184582
Title: Physical Exercise During Neoadjuvant Chemotherapy for Breast Cancer as a Means to Increase Pathological Complete Response Rates: the Randomized Neo-ACT Trial
Brief Title: Physical Exercise During Preoperative Chemotherapy for Breast Cancer
Acronym: Neo-ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jana de Boniface, Ass. Prof, PI, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo-ACT
Record Dates: First submitted 2021-12-07; First posted 2022-01-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: Randomization to supervised high-intensity interval training during neoadjuvant chemotherapy or usual information about physical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (No Intervention): Routine information on the benefit of physical activity
- Intervention (Experimental): High-intensity interval and strength training during neoadjuvant chemotherapy
  Interventions: Behavioral: Physical training

INTERVENTIONS:
Behavioral: Physical training — Participants randomized to the exercise group will complete two structured 60-min exercise sessions per week from initiation of NACT to surgery (approx. five months).
  Arms: Intervention

SUMMARY:
Neoadjuvant chemotherapy (NACT) is increasingly used in breast cancer. The best proof of NACT efficacy is pathological complete response (pCR), i.e. the absence of invasive tumour on post-NACT surgical histopathology. While it is known that physical exercise can help patients to better tolerate and complete often harsh cancer treatments, it is an emerging area of research to understand if and how exercise exerts anti-tumour effects and improves oncological outcomes.

The main aim of the Neo-ACT trial is to examine if a physical exercise intervention during NACT can increase pCR rates in breast cancer. Secondary aims are residual cancer burden, radiological tumour response, patient-related outcomes (health-related quality of life, physical activity), physiological outcomes (muscle strength, cardiorespiratory fitness), cancer treatment-related toxicities (cognitive dysfunction, chemotherapy completion rates) and long-term sick leave. Furthermore, the trial will explore how physical exercise affects anti-tumoral mechanisms inherent to therapy or host by hypothesis-generating translational analyses.

712 patients with primary invasive breast cancer will be randomized to either a supervised intervention of high-intensity interval and resistance training during NACT, supported by an exercise app, or to usual care, and followed for two years. Physical activity is meticulously tracked. By offering patients active involvement, the trial contributes strongly to the concept of personalized medicine.

DETAILED DESCRIPTION:
The Neo-ACT assesses the primary endpoint pathological complete response (pCR) and the secondary endpoints Residual Cancer Burden (RCB), objective tumour response (RECIST), all-cause, breast cancer-specific, and recurrence-free survival at 2, 5 and 10 years, health-related quality of life assessed by the EORTC QLQ-C30 and BR23 questionnaires, self-reported physical activity (Modified Godin Leisure Time Physical activity questionnaire), toxicity-related outcomes (chemotherapy completion rates, number of unplanned hospital admissions during NACT, objective cognitive dysfunction (Amsterdam Cognition Scan), cardiac toxicity and sick leave), device-measured physical activity level (Fitbit activity tracker), muscle strength (handgrip strength test and hypothetical 1-RM maximal leg muscle strength tests), and cardiorespiratory fitness (Ekblom-Bak submaximal cycle test).

Participants randomized to the exercise group will complete 120 min exercise sessions per week from initiation of NACT to surgery (approx. five months):

* Progressive home exercise program by an individualised mobile phone application, supported by local physiotherapists
* Initial exercise intensity individually tailored to each patient's fitness at baseline and rate of perceived exertion during the program and adapted if required
* Sessions will begin with a 3-minute moderate intensity (12-13 on Borg's Rate of Perceived Exertion (RPE) scale) warm-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary invasive breast cancer cT1-T3 cN0-2
* Full tumour biology available before initiation of NACT
* Oral and written consent
* Age ≥ 18 years

Exclusion Criteria:

* Pregnancy or breast-feeding
* Bilateral invasive breast cancer
* The presence of musculoskeletal, neurological, respiratory, metabolic or cardiovascular conditions that may prevent safe completion of the exercise demands of the study
* Currently performing equal to or more than 150 mins of moderate to high intensity aerobic exercise and 2 sessions per week of moderate intensity resistance exercise

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 5-6 months
  Absence of residual invasive tumor in breast and axilla at surgery

SECONDARY OUTCOMES:
Global health-related quality of life | baseline, after 1 and 2 years
  assessed by the EORTC QLQ-C30 questionnaire
Breast cancer-related quality of life | baseline, after 1 and 2 years
  assessed by the EORTC QLQ-B23 questionnaire
Self-reported physical activity | baseline, pre-surgery, 1- and 2-year follow-up
  Modified Godin Leisure Time Physical activity questionnaire
Chemotherapy completion rate | 1 year
  proportion of participants receiving the planned number of treatments
Cumulative chemotherapy dosage | 1 year
  total dose of NACT received to account for potential dose reduction
Objective cognitive dysfunction | baseline and 1 year
  online neuropsychological test (Amsterdam Cognition Scan)
Sick leave | pre-surgery and at 1- and 2-year follow-up
  Patient-reported absence from work
Device-measured physical activity level | baseline and 5-6months (pre surgery)
  Fit-bit tracker
Muscle strength | baseline and 5-6 months
  hypothetical 1-RM maximal leg muscle strength test
Handgrip strength | baseline and 5-6 months
  handgrip strength test
Cardiorespiratory fitness | baseline and 5-6 months (pre-surgery)
  Åstrand submaximal cycle test
Radiological tumour response | 5-6 months
  RECIST
Residual Cancer Burden (RCB) | 5-6 months
  Degree of tumor response to NACT

CONTACTS AND LOCATIONS:
Overall Officials: Jana de Boniface, Principal Investigator — Karolinska Institutet
Locations (13):
- Cabrini Health, Melbourne, Australia
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- Sweden (8):
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg
  - Skaraborgs sjukhus, Lidköping
  - Capio St Görans Hospital, Stockholm
  - Southern General Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Umeå University Hospital, Umeå
  - Västmanlands Hospital, Västerås
- United Kingdom (2):
  - Edinburgh Napier University, Edinburgh, Scotland
  - Royal Marsden, London

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available after study completion upon reasonable request submitted to the PI and with all legal and ethical requirements being fulfilled.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol, SAP and ICF available on trial homepage presently. Open access. CSR and analytic code available on request, see above.
URL: https://ki.se/en/mmk/the-neo-act-trial

REFERENCES:
- [Derived] de Boniface J, Altena R, Haddad Ringborg C, Bolam KA, Wengstrom Y. Physical exercise during neoadjuvant chemotherapy for breast cancer as a mean to increase pathological complete response rates: Trial protocol of the randomized Neo-ACT trial. PLoS One. 2022 Oct 13;17(10):e0274804. doi: 10.1371/journal.pone.0274804. eCollection 2022. PMID 36227931